CLINICAL TRIAL: NCT02505373
Title: A Novel Brief Therapy for Attempted Suicide: Two Year Follow-Up Randomized Controlled Study of the Attempted Suicide Short Intervention Program (ASSIP)
Brief Title: ASSIP, Attempted Suicide Short Intervention Program. Two Year Follow-Up Study
Acronym: ASSIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 144/08
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Suicide Attempt; Suicide; Suicidal Ideation
Keywords: Brief Therapy; Attempted Suicide; Therapeutic Alliance; Suicidal Ideation; Suicide; ASSIP
MeSH Terms: conditions — Suicide, Attempted; Suicide; Suicidal Ideation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group ASSIP (Experimental): Intervention Group ASSIP (Brief Therapy)
  Interventions: Behavioral: Attempted Suicide Short Intervention Program (ASSIP)
- Control Group CG (Active Comparator): Control Group CG (structured interview)
  Interventions: Behavioral: Control Group (CG)

INTERVENTIONS:
Behavioral: Attempted Suicide Short Intervention Program (ASSIP) — The brief therapy ASSIP consists of three to four sessions, which are ideally administered within a period of 2 to 4 weeks. Therapy sessions are scheduled for 60 to 90 minutes.
  Session 1: A narrative interview is conducted, in which the patient is asked to tell his or her personal story which led to the suicidal crisis. The narrative is video-recorded.
  Session 2: Using video-playback of the recorded narrative, patient and therapist explore further details of the suicidal process.
  Session 3: A case conceptualization focusing on the patient's vulnerability and the trigger of the suicidal crisis is formulated in writing. A list of safety strategies for the prevention of future suicidal behaviour is developed jointly with the patient.
  Regular letters are sent to patients over a period of 2 years.
  Arms: Intervention Group ASSIP
Behavioral: Control Group (CG) — Participants assigned to the control group underwent a single clinical interview that included a structured assessment of suicide using the SSF (Jobes, 2006).
  Arms: Control Group CG

SUMMARY:
Objective

Attempted suicide is the main risk factor for repeated suicidal behavior. However, evidence of the effectiveness of follow-up treatments for these patients is limited. The authors evaluated the effectiveness of the Attempted Suicide Short Intervention Program (ASSIP), a novel brief therapy based on a patient-oriented model of suicidal behavior. The ASSIP consists of three sessions followed by regular letters for 24 months.

Method

In this treatment study, 120 patients were randomly assigned to either the ASSIP intervention or a control group that received a one-session clinical assessment. Both groups received in- and outpatient treatment as usual. Study participants also completed a set of psychosocial and clinical questionnaires every 6 months during a 24-month follow-up period.

DETAILED DESCRIPTION:
Background

In the prevention and treatment of suicidality the main emphasis according to the traditional medical model has been on diagnosis and treatment of mental disorders, first and foremost depression. However, it is debatable how far this approach toward the suicidal patient can actually affect suicide rates. It has been argued that the mechanisms of suicidal behavior should be studied independently of any associated psychiatric disorder.

Follow-up studies strongly suggest that when a person has attempted suicide, the risk of future suicidal behavior, including death by suicide, cannot be "cured". Once a person has tried to solve an emotional crisis with a suicide attempt, this behavioral pattern will quickly re-emerge in similar situations in the future, not only because a suicide attempt provides a - temporary - solution, but also because very often it associated with an immediate sense of relief. The prevailing view emerging from recent developments in suicide research is that, following attempted suicide, it is crucial to establish individual safety strategies with patients for coping differently in future emotional crises. For as many patients as possible to benefit, treatments targeting suicidality should be brief and focused, and, of course, effective.

ASSIP combines aspects of action theory, cognitive behavior therapy, and attachment theory. A fundamental assumption is that an action theoretical approach toward the suicidal patient will establish a therapeutic alliance in the sense of a "secure base", which will enhance the effect of the regular letters following the four treatment sessions. ASSIP is not a stand-alone therapy but should be offered to suicidal patients in addition to the usual clinical management and follow-up treatment.

Objective

1. How effective is ASSIP, compared to a control group in preventing suicidal behaviour after a suicide attempt?

   1. Primary outcome measures: Suicidal behaviour, suicidal ideation
   2. Secondary outcome measures: Depression, coping skills, contact to health care system
2. Which parameters have a moderating influence on outcome measures?

   1. Therapeutic alliance
   2. Diagnosis
   3. Previous suicide attempts

Methods

In this treatment study, 120 patients were randomly assigned to either the ASSIP intervention or a control group that received a one-session clinical assessment. Both groups received in- and outpatient treatment as usual. The quality of the therapeutic alliance as a moderating factor for outcome was measured at the therapy sessions 1 (both groups) and 3 (ASSIP group only) using the Helping Alliance Questionnaire (HAq). Regarding outcome measures the study participants completed a set of psychosocial and clinical questionnaires every 6 months during a 24-months follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male/female
* Inpatient/outpatient, day care treatment
* German language
* All diagnosis (except: psychosis)
* Written informed consent

Exclusion Criteria

* Psychosis
* Imprisonment
* Foreign languages

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Suicidal behaviour | 2-year follow-up
  Measured by socio-demographic & clinical questionnaire
Suicidal behaviour | 1-year follow-up
  Measured by socio-demographic & clinical questionnaire

SECONDARY OUTCOMES:
Contact to health care system | At baseline, after 6 months, after 12 months, after 18 months, after 24 months
  Measured by questionnaire
Suicidal ideation | At baseline, after 6 months, after 12 months, after 18 months, after 24 months
  Measured by Beck Scale for Suicidal Ideation (BSS)
Depression | At baseline, after 6 months, after 12 months, after 18 months, after 24 months
  Measured by Beck Depression Inventory (BDI)
Coping | At baseline, after 6 months, after 12 months, after 18 months, after 24 months
  Measured by Brief COPE
Global distress | At baseline, after 6 months, after 12 months, after 18 months, after 24 months
  Measured by SCL-9

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Michel, Prof., Principal Investigator — Hospital of Psychiatry and Psychotherapy, University of Bern; Anja C Gysin-Maillart, Ph.D., Principal Investigator — Hospital of Psychiatry and Psychotherapy, University of Bern
Locations (1):
- University Hospital of Psychiatry and Psychotherapy, University of Bern, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Alexander, L. B. & Luborsky, L. (1986).The Penn Helping Alliance Scales. In L. S. Greenberg & W. M. Pinsoff (Eds.), The psychotherapeutic process: A research handbook (pp. 325-366). New York, NY: Guilford Press.
- [Background] Arensman E, Townsend E, Hawton K, Bremner S, Feldman E, Goldney R, Gunnell D, Hazell P, Van Heeringen K, House A, Owens D, Sakinofsky I, Traskman-Bendz L. Psychosocial and pharmacological treatment of patients following deliberate self-harm: the methodological issues involved in evaluating effectiveness. Suicide Life Threat Behav. 2001 Summer;31(2):169-80. doi: 10.1521/suli.31.2.169.21516. PMID 11459249
- [Background] Beck, A. T. & Steer, R. A. (1987). BDI, Beck depression inventory: manual. New York, NY: Psychological Corporation.
- [Background] Beck, A. T. & Steer, R. A. (1991). Manual for the Beck scale for suicide ideation. San Antonio, TX: Psychological Corporation.
- [Background] Brown GK, Ten Have T, Henriques GR, Xie SX, Hollander JE, Beck AT. Cognitive therapy for the prevention of suicide attempts: a randomized controlled trial. JAMA. 2005 Aug 3;294(5):563-70. doi: 10.1001/jama.294.5.563. PMID 16077050
- [Background] Carter GL, Clover K, Whyte IM, Dawson AH, D'Este C. Postcards from the EDge: 5-year outcomes of a randomised controlled trial for hospital-treated self-poisoning. Br J Psychiatry. 2013 May;202(5):372-80. doi: 10.1192/bjp.bp.112.112664. Epub 2013 Mar 21. PMID 23520223
- [Background] Claassen CA, Pearson JL, Khodyakov D, Satow PM, Gebbia R, Berman AL, Reidenberg DJ, Feldman S, Molock S, Carras MC, Lento RM, Sherrill J, Pringle B, Dalal S, Insel TR. Reducing the burden of suicide in the U.S.: the aspirational research goals of the National Action Alliance for Suicide Prevention Research Prioritization Task Force. Am J Prev Med. 2014 Sep;47(3):309-14. doi: 10.1016/j.amepre.2014.01.004. Epub 2014 Apr 18. PMID 24750971
- [Background] Granboulan V, Roudot-Thoraval F, Lemerle S, Alvin P. Predictive factors of post-discharge follow-up care among adolescent suicide attempters. Acta Psychiatr Scand. 2001 Jul;104(1):31-6. doi: 10.1034/j.1600-0447.2001.00297.x. PMID 11437747
- [Background] Gysin-Maillart, A. & Michel, K. (2013). Kurztherapie nach Suizidversuch. ASSIP-Attempted Suicide Short Intervention Program. Therapiemanual. Bern: Huber. ISBN: 9783456852386
- [Background] Hatcher S, Sharon C, Coggan C. Beyond randomized controlled trials in attempted suicide research. Suicide Life Threat Behav. 2009 Aug;39(4):396-407. doi: 10.1521/suli.2009.39.4.396. PMID 19792981
- [Background] Jobes DA. Collaborating to prevent suicide: a clinical-research perspective. Suicide Life Threat Behav. 2000 Spring;30(1):8-17. PMID 10782715
- [Background] Monti, K., Cedereke, M. & Ojehagen, A. (2003). Treatment attendance and suicidal behavior 1 month and 3 months after a suicide attempt: A comparison between two samples. Archives of Suicide Research, 7, 167-174. http://doi.org/10.1080/13811110301581
- [Background] Michel, K. & Valach, L. (1997). Suicide as goal-directed action. Archives of Suicide Research, 3, 213-221. http://doi.org/10.1080/13811119708258273
- [Background] Michel K, Dey P, Stadler K, Valach L. Therapist sensitivity towards emotional life-career issues and the working alliance with suicide attempters. Arch Suicide Res. 2004;8(3):203-13. doi: 10.1080/13811110490436792. PMID 16081387
- [Background] Michel K, Maltsberger JT, Jobes DA, Leenaars AA, Orbach I, Stadler K, Dey P, Young RA, Valach L. Discovering the truth in attempted suicide. Am J Psychother. 2002;56(3):424-37. doi: 10.1176/appi.psychotherapy.2002.56.3.424. PMID 12400207
- [Background] Michel, K. & Gysin-Maillart, A. (2015). Attempted Suicide Short Intervention Program ASSIP. A manual for clinicians. Göttingen: Hogrefe. ISBN: 978-0-88937-476-8
- [Background] Motto JA, Bostrom AG. A randomized controlled trial of postcrisis suicide prevention. Psychiatr Serv. 2001 Jun;52(6):828-33. doi: 10.1176/appi.ps.52.6.828. PMID 11376235
- [Background] Rudd MD, Bryan CJ, Wertenberger EG, Peterson AL, Young-McCaughan S, Mintz J, Williams SR, Arne KA, Breitbach J, Delano K, Wilkinson E, Bruce TO. Brief cognitive-behavioral therapy effects on post-treatment suicide attempts in a military sample: results of a randomized clinical trial with 2-year follow-up. Am J Psychiatry. 2015 May;172(5):441-9. doi: 10.1176/appi.ajp.2014.14070843. Epub 2015 Feb 13. PMID 25677353
- [Background] Rudd MD. The suicidal mode: a cognitive-behavioral model of suicidality. Suicide Life Threat Behav. 2000 Spring;30(1):18-33. PMID 10782716
- [Background] Silverman MM, Berman AL, Sanddal ND, O'carroll PW, Joiner TE. Rebuilding the tower of Babel: a revised nomenclature for the study of suicide and suicidal behaviors. Part 2: Suicide-related ideations, communications, and behaviors. Suicide Life Threat Behav. 2007 Jun;37(3):264-77. doi: 10.1521/suli.2007.37.3.264. No abstract available. PMID 17579539
- [Background] Stanley, B. & Brown, G. K. (2012). Safety planning intervention: A brief intervention to mitigate suicide risk. Cognitive and Behavioral Practice, 19, 256-264. http://doi.org/10.1016/j.cbpra.2011.01.001
- [Background] Zelen M. A new design for randomized clinical trials. N Engl J Med. 1979 May 31;300(22):1242-5. doi: 10.1056/NEJM197905313002203. PMID 431682
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Gibbon S, Khalifa NR, Cheung NH, Vollm BA, McCarthy L. Psychological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007668. doi: 10.1002/14651858.CD007668.pub3. PMID 32880104
- [Derived] Park AL, Gysin-Maillart A, Muller TJ, Exadaktylos A, Michel K. Cost-effectiveness of a Brief Structured Intervention Program Aimed at Preventing Repeat Suicide Attempts Among Those Who Previously Attempted Suicide: A Secondary Analysis of the ASSIP Randomized Clinical Trial. JAMA Netw Open. 2018 Oct 5;1(6):e183680. doi: 10.1001/jamanetworkopen.2018.3680. PMID 30646253
- [Derived] Gysin-Maillart A, Schwab S, Soravia L, Megert M, Michel K. A Novel Brief Therapy for Patients Who Attempt Suicide: A 24-months Follow-Up Randomized Controlled Study of the Attempted Suicide Short Intervention Program (ASSIP). PLoS Med. 2016 Mar 1;13(3):e1001968. doi: 10.1371/journal.pmed.1001968. eCollection 2016 Mar. PMID 26930055